CLINICAL TRIAL: NCT02962245
Title: Efficacy of Treatment With Berberine to Maintain Remission in Ulcerative Colitis: An Open-label,Randomized,Phase IV Clinical Trial
Brief Title: Efficacy of Treatment With Berberine to Maintain Remission in Ulcerative Colitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20162062-1
Record Dates: First submitted 2016-10-14; First posted 2016-11-11 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Berberine
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Berberine

ARMS (2):
- berberine group (Active Comparator): regular treatment and receive oral berberine 300mg three times daily untill recurrence in one year
  Interventions: Drug: berberine; Drug: regular treatment
- regular treatment group (Placebo Comparator): regular treatment untill recurrence in one year
  Interventions: Drug: regular treatment

INTERVENTIONS:
Drug: berberine
  Arms: berberine group
Drug: regular treatment — such as 5-ASA,immunomodulating/suppressive agents or Anti-TNF therapy

SUMMARY:
The research aim to find out whether berberine can reduce the annual recurrence rate of ulcerative colitis in remission.

A total of 238 patients with ulcerative colitis in remission will be randomly divided into two groups.One will receive regular treatment,and the other group will receive extra oral berberine 300 mg three times daily for a year.

The end of the study for every patient is disease recurrence(Mayo Clinic score of 3 points or more ).

The primary analysis is annual recurrence rate, and both endoscopy and Mayo Clinic disease activity index scores at the baseline and final assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with ulcerative colitis(according to the second European evidence-based consensus on the diagnosis and management of ulcerative colitis);
2. Disease remission of ulcerative colitis(a total Mayo Clinic score of 2 points or less and an endoscopic score of 1 point or less);
3. Diagnosis of moderate or severe ulcerative colitis within 3 months(a total Mayo Clinic score of 6-12 points)

Exclusion Criteria:

1. Prior bowel resection surgery;
2. Women who are planning or actual pregnancy or lactation during study period;
3. Patients allergic to berberine;
4. History of disease that would interfere with their participation in the trial, including malignant diseases, bleeding disorders, active gastric or active duodenal ulcers, autoimmune diseases, and mental or emotional disorder;
5. Take the following treatment:

   * Unstable dose of 5-ASA drugs (oral and/or rectal route) within 14 days prior to screening;
   * Unstable dose of any immunomodulating/suppressive agents and any Anti-TNF therapy within 3 months prior to screening;
   * Traditional Chinese Medicine for the treatment of UC (any pharmaceutical form) within 7 days prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Annual Recurrence Rate | a year

SECONDARY OUTCOMES:
Disease exacerbation rate measured by Mayo Clinic disease activity index scores | a year
  The primary analysis is disease exacerbation through day 14 among patients who underwent randomization, had Mayo Clinic disease activity index scores at the baseline and final assessments. Disease exacerbation is defined as a total Mayo Clinic score of 5 points or more and an increase in the endoscopic score of 1 point or more.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | a year